CLINICAL TRIAL: NCT04156893
Title: RH Genotype Matched Red Cell Transfusions for Patients With Sickle Cell Disease
Brief Title: RH Genotype Matched RBC Transfusions
Acronym: RBC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: New York Blood Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-016565; R01HL147879 (NIH); R01HL169401 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cells Disease
Keywords: Chronic Transfusion

STUDY DESIGN:
Intervention Model Description: Subjects will receive RH genotype matched red cell units for transfusion. For subjects with a history of stroke/recurrent transient ischemic attack or other indication who require tight control of Hb S, and RH genotyped blood is not available, standard of care serologic matched blood would be administered rather than delaying transfusion and risking higher Hb S level.
  For all subjects, standard of care serologic matched blood would be administered rather than delaying transfusion beyond 7 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RH genotype matched red cell transfusions (Experimental): Subjects will receive RH genotyped matched red cell units for transfusion in addition to standard serologic C, E, and K antigen matching and being hemoglobin S negative, which is our institutional standard of care for patients with Sickle Cell Disease.
  Interventions: Biological: Red cell units that are genotype matched at the RHD and RHCE loci

INTERVENTIONS:
Biological: Red cell units that are genotype matched at the RHD and RHCE loci — Patients will be provided with red cell units that are C, E, and K antigen matched (standard of care for patients with SCD) and genotype matched at the RHD and RHCE loci.

SUMMARY:
To determine the feasibility and efficacy of matching donor red cells by RH genotype for a cohort of chronically transfused patients with SCD.

DETAILED DESCRIPTION:
This is a Phase 1/2 trial in patients with Sickle Cell Disease requiring chronic red cell transfusions. RH genotyped donor units will be obtained from the New York Blood Center. Patients will be matched with donor units whose RH genotypes predict no foreign Rh protein exposure to the patient. This will provide red cell matching at a level above the current standard of care (serologic C, E, and K matching). Patients will receive RH matched red cells for the duration of their chronic transfusion therapy or up to three years, whichever is shorter. In the pilot phase, we have determined it is feasible to identify RH matched donor units for the patient's RH genotype for every scheduled transfusion. We will now continue to show feasibility as well as determine efficacy by monitoring Rh alloantibody formation.

For subjects with a history of stroke/recurrent transient ischemic attack or other indication who require tight control of Hb S, and RH genotyped blood is not available, standard of care serologic matched blood would be administered rather than delaying transfusion and risking higher Hb S level.

For all subjects, standard of care serologic matched blood would be administered rather than delaying transfusion beyond 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age >6 months
* Diagnosis of SCD, all genotypes
* Require a period of chronic red cell transfusion therapy
* Subject/parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria:

* Rare RH genotype that would preclude identification of sufficient RBC units
* Antigen negative requirements due to alloimmunization that would preclude identification of sufficient RBC units
* Alloimmunized to D antigen
* Rh alloimmunized patients for whom providing RH genotype matched blood would expose the patient to an antigen that would not be consistent with standard of care and blood bank protocols
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Determine the treatment efficacy by monitoring the rate of Rh alloimmunization | 3.5 years
  A primary objective is to determine whether providing RH genotype matched red cell units can reduce or prevent Rh alloimmunization.
Determine the feasibility of identifying sufficient RH genotype matched units | 3.5 years
  A primary objective is to determine the feasibility of identifying sufficient RH genotype matched red cells for chronically transfused patients with SCD with varied RH genotypes. Approximately 20 RHD (Rhesus D) and 20 RHCE (Rhesus CE) variants have been observed in patients with SCD and will determine whether sufficient RH genotyped units can be matched to the patient's own RH genotype.

SECONDARY OUTCOMES:
Determine the rate of non-Rh alloimmunization | 3.5 years
  A secondary objective is to determine the rate of antibody formation outside the Rh blood group system, such as anti-Kidd or -S/s.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Chou, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Protected Health Information (PHI) will be shared with the New York Blood Center (NYBC) to order blood for the subjects. This will be done using a secure online blood ordering system. The NYBC uses an FDA-approved HIPAA secure system called Blood Enterprise Computer System (BECS) to store patient data and results, including PHI. 3rd party computers at New York Blood Center will also store study data using study identification (ID) numbers. The purpose of having study data coded at NYBC is for specialized testing for red antigens or antibodies for which we will provide some clinical data to assist in the laboratory evaluation. To assure that the transmission of data and samples maintains confidentiality we will used study ID numbers for these samples. The master list will be maintained at the Children's Hospital of Philadelphia (CHOP). The study databases are password protected and on password protected computers at CHOP and at NYBC, that are backed up on the research servers.
Supporting Information: Study Protocol
Time Frame: For the duration of the study
Access Criteria: Only study team members will have access to the data.

REFERENCES:
- [Background] Chou ST, Jackson T, Vege S, Smith-Whitley K, Friedman DF, Westhoff CM. High prevalence of red blood cell alloimmunization in sickle cell disease despite transfusion from Rh-matched minority donors. Blood. 2013 Aug 8;122(6):1062-71. doi: 10.1182/blood-2013-03-490623. Epub 2013 May 30. PMID 23723452
- [Background] Vichinsky EP, Earles A, Johnson RA, Hoag MS, Williams A, Lubin B. Alloimmunization in sickle cell anemia and transfusion of racially unmatched blood. N Engl J Med. 1990 Jun 7;322(23):1617-21. doi: 10.1056/NEJM199006073222301. PMID 2342522
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Chou ST, Evans P, Vege S, Coleman SL, Friedman DF, Keller M, Westhoff CM. RH genotype matching for transfusion support in sickle cell disease. Blood. 2018 Sep 13;132(11):1198-1207. doi: 10.1182/blood-2018-05-851360. Epub 2018 Jul 19. PMID 30026182
- [Background] Coleman S, Westhoff CM, Friedman DF, Chou ST. Alloimmunization in patients with sickle cell disease and underrecognition of accompanying delayed hemolytic transfusion reactions. Transfusion. 2019 Jul;59(7):2282-2291. doi: 10.1111/trf.15328. Epub 2019 Apr 25. PMID 31021439